CLINICAL TRIAL: NCT07004777
Title: Effect of Consuming n-3 Polyunsaturated Fatty Acids Rich Foods on Triglyceride Concentration and Lipoprotein Composition in Individuals With Hypertriglyceridemia. Controlled Clinical Trial.
Brief Title: Effect of Consuming n-3 PUFAs Rich Foods on Triglyceride Concentration and Lipoprotein Composition
Acronym: SALVIMEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Martha Guevara Cruz, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNU-5515-25-27-1; INCMNSZ (Other: INCMNSZ)
Record Dates: First submitted 2025-05-20; First posted 2025-06-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia; Lipid metabolism; Dyslipidemia; Fatty Acids, Omega-3; Eicosapentaenoic Acid; Docosahexaenoic Acid; diet
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: The groups will receive the treatment simultaneously.
Who Masked: Outcomes Assessor
Masking Description: The person who will perform the biochemical determinations and the statistical analysis will be blinded from the intervention group by assigning each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Salmon diet (Experimental): Diet based on participant-specific energy expenditure. With the following macronutrient distribution: 50% carbohydrates, protein 20% and 30% fats.
  Interventions: Other: Isocaloric diet including salmon
- Chia and pumpkin seeds diet (Experimental): Diet based on participant-specific energy expenditure. With the following macronutrient distribution: 50% carbohydrates, protein 20% and 30% fats.
  Interventions: Other: Isocaloric diet including chia and pumpkin seeds
- Diet plus fish oil (Active Comparator): Diet based on participant-specific energy expenditure. With the following macronutrient distribution: 50% carbohydrates, protein 20% and 30% fats.
  Interventions: Dietary Supplement: Isocaloric diet plus fish oil

INTERVENTIONS:
Other: Isocaloric diet including chia and pumpkin seeds — Diet based on participant-specific energy expenditure. With the following macronutrient distribution: 50% carbohydrates, protein 20% and 30% fats.
  This dietary intervention consists of a four-week follow-up period and incorporates the intake of pumpkin and chia seeds.
  Arms: Chia and pumpkin seeds diet
Dietary Supplement: Isocaloric diet plus fish oil — Diet based on participant-specific energy expenditure. With the following macronutrient distribution: 50% carbohydrates, protein 20% and 30% fats.
  This dietary intervention consists of a four-week follow-up period and incorporates EPA + DHA supplement (fish oil) to the diet.
  Arms: Diet plus fish oil
Other: Isocaloric diet including salmon — Diet based on participant-specific energy expenditure. With the following macronutrient distribution: 50% carbohydrates, protein 20% and 30% fats.
  This dietary intervention consists of a four-week follow-up period and incorporates the intake of salmon.
  Arms: Salmon diet

SUMMARY:
Hypertriglyceridemia is one of the most prevalent lipid profile disorders and is linked to a large proportion of mortality in Mexico and around the world. Various international treatment guidelines for hypertriglyceridemia have suggested the consumption of foods rich in n-3 polyunsaturated fatty acids or their intake through supplementation as a complement to lifestyle changes. However, adherence to the consumption of foods and supplements containing these fatty acids is often limited due to lack of acceptance or unaffordability. For this reason the objective of the study is to evaluate the effect and adherence to the consumption of foods rich in n-3 polyunsaturated fatty acids (PUFA) (pumpkin and chia seeds and salmon) and n-3 PUFA supplement during four weeks of a follow up dietary intervention determined by triglyceride concentration and lipoprotein composition in people with hypertriglyceridemia.

The study is divided into two phases. In the first, participants' diets will be standardized, providing them with dietary recommendations for four weeks.

Participants who maintain triglyceride levels >200 mg/dL despite the recommendations will be invited to a second phase: a randomized controlled clinical trial consisting of a dietary intervention with a four-week follow-up.

Participants will be randomized into three treatment groups: 1) isocaloric diet and Eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA) supplementation; 2) isocaloric diet including salmon; 3) isocaloric diet including chia and pumpkin seeds. The effect of the dietary intervention will be assessed by determining lipid composition and lipoprotein analysis, while adherence to n-3 PUFA consumption will be measured by serum fatty acid profile analysis.

DETAILED DESCRIPTION:
The study is divided into two phases. The first phase is a prospective study with a 4-week follow-up to standardize the participants' diet. The second phase is a randomized controlled clinical trial consisting of a dietary intervention with a four-week follow-up.

Phase 1

Participants' diets will be standardized using dietary recommendations based on guidelines. Individuals who agree to participate will be required to sign an informed consent form. At baseline and at the end of this phase, participants will undergo a medical history questionaire, anthropometric assessments (weight, height, and waist circumference), body composition analysis (body fat percentage, skeletal muscle mass percentage, and lean muscle mass percentage), blood pressure measurement, and cardiometabolic risk score evaluation. Additionally, blood samples will be collected to determine serum concentrations of glucose, lipid profile parameters (total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, and triglycerides) as well as for the isolation of monocytes to determine mitochondrial function. It will be recommended to the participants to continue with the dietary recommendations until transitioning to the clinical trial, where those whose triglyceride concentrations remain >200 mg/dL will be invited to participate.

Phase 2

Participants with hypertriglyceridemia will be randomly assigned to three groups, each of which will be prescribed an isocaloric diet including a food or supplement rich in n-3 PUFA:

* An isocaloric diet and EPA+DHA supplement
* An isocaloric diet including salmon
* An isocaloric diet including chia seeds

Resting energy expenditure wil be measured by indirect calorimetry to determine energy requirement of each participant. Distribution of micronutrients of the dietary intervention will be as follow: 50% carbohydrates, 20% protein, and 30% lipids .

This dietary intervention will last 4 weeks. To promote adherence, participants will be given foods or supplements rich in n-3 PUFA.

The same assessments conducted in the previous phase will be repeated at the start and at the end of the 4 week-follow-up period of the intervention. Additionally, other parameters will be evaluated, including insulin levels; inflammatory markers ; endothelial markers and intercellular adhesion molecule-1, cardiometabolic risk markers ; oxidative stress markers; liver function tests ; and pulse wave velocity. Lipid composition and lipoprotein analysis will also be determined to evaluate the effect. As well as the concentration of serum fatty acid profile analysis to evaluate the adherence to PUFA-n3.

In both phases, dietary intake and the adherence to dietary treatment will be monitored using 24-hour dietary recalls, which will be conducted during all visits, as well as through phone calls 2 times per week and text messages.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Signing of the informed consent form
* Both sexes.
* Adults over 18 years of age.
* BMI >18.5 kg/m2.
* Triglycerides between 200 and 500 mg/dL.
* Total cholesterol less than 240 mg/dL

Phase 2

* Both sexes
* Adults over 18 years of age.
* BMI >18.5 kg/m2
* Individuals whose triglyceride concentration is greater than 200 mg/dL and less than 500 mg/dL after dietary treatment (dietary recommendations based on the National Cholesterol Education Program - Adult Treatment Panel III (NCEP-ATPIII) guidelines).

Exclusion Criteria:

* Any type of diabetes.
* kidney disease diagnosed by a physician.
* Acquired diseases that secondarily cause obesity and diabetes.
* Patients who have suffered a cardiovascular event.
* Weight loss >3 kg in the last 3 months.
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Pregnancy.
* Treatment with any medication:
* Treatment with antihypertensive drugs (tricyclic, loop, or potassium-sparing diuretics, angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, alpha-blockers, calcium channel blockers, beta-blockers).
* Treatment with hypoglycemic agents (sulfonylureas, biguanides, incretins) or - insulin and antidiabetics.
* Treatment with statins, fibrates, or other drugs to control dyslipidemia.
* Use of steroid medications, chemotherapy, immunosuppressants, or radiation therapy.
* Anorectic agents or those that accelerate weight loss.
* Treatment with any medication that influences inflammation (corticosteroids, nonsteroidal anti-inflammatory drugs, colchicine, interleukin-1 inhibitors) or triglyceride metabolism (metformin, glitazones, SGLT2 inhibitors, fibrates, statins, cholesterol ester transporter protein (CETP) inhibitors, pancreatic lipase inhibitors).
* Anticoagulants and antiplatelets (warfarin, aspirin, clopidogrel).
* People with a smoking cessation index (SCI) greater than 21.
* People with a tobacco Index greater than 21.
* Consumption of large amounts of alcohol (14 drinks for women or 21 drinks for men in a typical week).
* Consumption of any recreational psychoactive substance.
* Allergy or intolerance to any food listed in the proposed pantry.
* Unwillingness to consume any of the foods listed in the proposed pantry.
* Previous n-3 PUFA supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum triglycerides concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum triglycerides between different nutrition interventions.
Serum fatty acid profile analysis by gas chromatography in microgram | From week 4 to week 8 of the intervention
  Change in serum fatty acid between different nutrition interventions.

SECONDARY OUTCOMES:
Serum total cholesterol concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum total cholesterol between different nutrition interventions.
Serum LDL cholesterol concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum LDL cholesterol between different nutrition interventions.
Serum HDL cholesterol concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum HDL cholesterol between different nutrition interventions.
Serum lipids concentration in relative peak area | From week 4 to week 8 of the intervention
  Change in serum lipids between different nutrition interventions.
Serum C-reactive protein concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum C-reactive protein between different nutrition interventions.
Plasma malondialdehyde concentration in nmol/mL | From week 4 to week 8 of the intervention
  Change in plasma malondialdehyde between different nutrition interventions.
Serum Intercellular Adhesion Molecule-1 (ICAM-1) concentration in pg/mL | From week 4 to week 8 of the intervention
  Change in serum ICAM-1 between different nutrition interventions.
Serum Vascular Cell Adhesion Molecule-1 (VCAM-1) concentration in pg/mL | From week 4 to week 8 of the intervention
  Change in serum VCAM-1 between different nutrition interventions.
Serum plasminogen concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum plasminogen between different nutrition interventions.
Serum glucose concentration in mg/dL | From week 4 to week 8 of the intervention
  Change in serum glucose between different nutrition interventions.
Serum aspartate aminotransferase concentration in IU/mL | From week 4 to week 8 of the intervention
  Change in serum aspartate aminotransferase between different nutrition interventions.
Serum alanine aminotransferase concentration in IU/mL | From week 4 to week 8 of the intervention
  Change in serum alanine aminotransferase between different nutrition interventions.
Serum insulin concentration in micro - IU / ml | From week 4 to week 8 of the intervention
  Change in serum insulin between different nutrition interventions.
Oxygen consumption rate in pmol of oxygen per minute per cell(s) | From week 4 to week 8 of the intervention
  Change in oxygen consumption rate between different nutrition interventions.
Body weight in kilograms | From week 4 to week 8 of the intervention
  Change in body weight between different nutrition interventions.
Waist circumference in centimeters | From week 4 to week 8 of the intervention
  Change in waist circumference between different nutrition interventions.
Fat mass percentage | From week 4 to week 8 of the intervention
  Change in fat mass percentage between different nutrition interventions.
Skeletal muscle mass percentage | From week 4 to week 8 of the intervention
  Change in skeletal muscle mass percentage between different nutrition interventions.
Lean mass percentage | From week 4 to week 8 of the intervention
  Change in lean mass percentage between different nutrition interventions.
Medium very low density lipoprotein (VLDL) particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma medium VLDL particle number between different nutrition interventions.
Large very low density lipoprotein (VLDL) particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma large VLDL particle number between different nutrition interventions.
Small very low density lipoprotein (VLDL) particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma small VLDL particle number between different nutrition interventions.
Large LDL particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma large LDL particle number between different nutrition interventions.
Medium LDL particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma medium LDL particle number between different nutrition interventions.
Small LDL particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma small LDL particle number between different nutrition interventions.
Large HDL particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma large HDL particle number between different nutrition interventions.
Small HDL particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma small HDL particle number between different nutrition interventions.
Medium HDL particle number in nmol/L | From week 4 to week 8 of the intervention
  Change in plasma medium HDL particle number between different nutrition interventions.
Pulse wave velocity in m/s | From week 4 to week 8 of the intervention
  Change in pulse wave velocity between different nutrition interventions
Controlled attenuation parameter in decibels per meter | From 4 week to 8 week of intervention
  Allows to evaluate the degree of steatosis by elastography.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Guevara, Study Director — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ly R, MacIntyre BC, Philips SM, McGlory C, Mutch DM, Britz-McKibbin P. Lipidomic studies reveal two specific circulating phosphatidylcholines as surrogate biomarkers of the omega-3 index. J Lipid Res. 2023 Nov;64(11):100445. doi: 10.1016/j.jlr.2023.100445. Epub 2023 Sep 18. PMID 37730162
- [Background] Ottestad I, Hassani S, Borge GI, Kohler A, Vogt G, Hyotylainen T, Oresic M, Bronner KW, Holven KB, Ulven SM, Myhrstad MC. Fish oil supplementation alters the plasma lipidomic profile and increases long-chain PUFAs of phospholipids and triglycerides in healthy subjects. PLoS One. 2012;7(8):e42550. doi: 10.1371/journal.pone.0042550. Epub 2012 Aug 28. PMID 22952598
- [Background] Erkkila AT, Manninen S, Fredrikson L, Bhalke M, Holopainen M, Ruuth M, Lankinen M, Kakela R, Oorni K, Schwab US. Lipidomic changes of LDL after consumption of Camelina sativa oil, fatty fish and lean fish in subjects with impaired glucose metabolism-A randomized controlled trial. J Clin Lipidol. 2021 Sep-Oct;15(5):743-751. doi: 10.1016/j.jacl.2021.08.060. Epub 2021 Sep 7. PMID 34548243
- [Background] Tatsuno I, Kudou K, Kagawa T. Effect of TAK-085 on Low-density Lipoprotein Particle Size in Patients with Hypertriglyceridemia: A Double-blind Randomized Clinical Study. Cardiovasc Ther. 2015 Dec;33(6):317-23. doi: 10.1111/1755-5922.12146. PMID 26222126
- [Background] Makni M, Fetoui H, Gargouri NK, Garoui el M, Jaber H, Makni J, Boudawara T, Zeghal N. Hypolipidemic and hepatoprotective effects of flax and pumpkin seed mixture rich in omega-3 and omega-6 fatty acids in hypercholesterolemic rats. Food Chem Toxicol. 2008 Dec;46(12):3714-20. doi: 10.1016/j.fct.2008.09.057. Epub 2008 Oct 1. PMID 18938206
- [Background] Avila-Nava A, Noriega LG, Tovar AR, Granados O, Perez-Cruz C, Pedraza-Chaverri J, Torres N. Food combination based on a pre-hispanic Mexican diet decreases metabolic and cognitive abnormalities and gut microbiota dysbiosis caused by a sucrose-enriched high-fat diet in rats. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201501023. Epub 2016 Aug 8. PMID 27352915
- [Background] Bhatt DL, Steg PG, Brinton EA, Jacobson TA, Miller M, Tardif JC, Ketchum SB, Doyle RT Jr, Murphy SA, Soni PN, Braeckman RA, Juliano RA, Ballantyne CM; REDUCE-IT Investigators. Rationale and design of REDUCE-IT: Reduction of Cardiovascular Events with Icosapent Ethyl-Intervention Trial. Clin Cardiol. 2017 Mar;40(3):138-148. doi: 10.1002/clc.22692. Epub 2017 Mar 15. PMID 28294373
- [Background] Zheng J, Huang T, Yu Y, Hu X, Yang B, Li D. Fish consumption and CHD mortality: an updated meta-analysis of seventeen cohort studies. Public Health Nutr. 2012 Apr;15(4):725-37. doi: 10.1017/S1368980011002254. Epub 2011 Sep 14. PMID 21914258
- [Background] Kontostathi M, Isou S, Mostratos D, Vasdekis V, Demertzis N, Kourounakis A, Vitsos A, Kyriazi M, Melissos D, Tsitouris C, Karalis E, Klamarias L, Dania F, Papaioannou GT, Roussis V, Polychronopoulos E, Anastassopoulou J, Theophanides T, Rallis MC, Black HS. Influence of Omega-3 Fatty Acid-Rich Fish Oils on Hyperlipidemia: Effect of Eel, Sardine, Trout, and Cod Oils on Hyperlipidemic Mice. J Med Food. 2021 Jul;24(7):749-755. doi: 10.1089/jmf.2020.0114. Epub 2020 Dec 23. PMID 33370175